CLINICAL TRIAL: NCT00004193
Title: Phase II Trial of ISIS 2503, an Antisense Inhibitor of H-ras, in Patients With Advanced Colorectal Cancer
Brief Title: ISIS 2503 in Treating Patients With Metastatic and/or Locally Recurrent Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067434; UAB-9860; ISIS-2503-CS6; NCI-G99-1649
Record Dates: First submitted 2000-01-21; First posted 2004-08-05 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — ISIS 2503

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ISIS 2503 (Experimental): patients who have metastatic and/or locally recurrent colorectal cancer
  Interventions: Drug: ISIS 2503

INTERVENTIONS:
Drug: ISIS 2503

SUMMARY:
RATIONALE: ISIS 2503 may kill cancer cells by inhibiting a gene that promotes the development and growth of cancer.

PURPOSE: Phase II trial to study the effectiveness of ISIS 2503 in treating patients who have metastatic and/or locally recurrent colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, duration of response, and time to progression in patients with metastatic and/or locally recurrent adenocarcinoma of the colon or rectum treated with ISIS 2503, an antisense inhibitor of H-ras. II. Determine the safety profile of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive ISIS 2503 IV continuously for 14 days. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic and/or locally recurrent adenocarcinoma of the colon or rectum that is not expected to be cured with standard therapy Patients who previously underwent definitive surgical resection and subsequently develop metastatic disease should have diagnosis reconfirmed with new histologic or cytologic specimen if: More than 5 years have elapsed since primary surgery OR Primary tumor was stage I or II At least 1 measurable lesion (2 cm or more in widest diameter) by CT or MRI scan No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0 or 1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dl Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study No underlying disease state associated with active bleeding No active infection requiring therapy No second malignancy within the past 5 years except curatively treated nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for metastatic disease At least 6 months since prior adjuvant chemotherapy with or without radiotherapy Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy to nonindicator lesion allowed and recovered See Chemotherapy Surgery: See Disease Characteristics Other: No concurrent approved cancer therapy or other experimental therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1999-01; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Determine the response rate, duration of response, and time to progression in patients with metastatic and/or locally recurrent adenocarcinoma of the colon or rectum treated with ISIS 2503, an antisense inhibitor of H-ras | baseline to survival

SECONDARY OUTCOMES:
Determine the safety profile of this regimen in these patients. | Baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor N. Saleh, MD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama Comprehensive Cancer Center, Birmingham, Alabama, United States